CLINICAL TRIAL: NCT01509027
Title: A Randomized Controlled Trial to Evaluate the Impact of Education on the Knowledge About and Compliance With a Phosphorus Restricted Diet and Phosphate Binder Therapy in Maintenance Dialysis Patients
Brief Title: Study of the Compliance With Phosphorus Restricted Diet and Phosphate Binder Therapy in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B322201112895
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Kidney Disease
Keywords: hemodialysis; hyperphoshatemia; compliance
MeSH Terms: conditions — Renal Insufficiency, Chronic; Patient Compliance | interventions — Standard of Care; Nutritionists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Education by DVD and dietician (Active Comparator): Information on detrimental conseqences of hyperphosphatemia is presented on DVD and individual dietary counseling is given by dieticican
  Interventions: Behavioral: Education by DVD and dietician
- Education by unpersonalised DVD (Active Comparator): Information on detrimental consequences of hyperphosphatemia is presented on DVD
  Interventions: Behavioral: education by DVD
- Standard Care (Placebo Comparator): standard care
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: education by DVD — Information on detrimental conseqences of hyperphosphatemia is presented on DVD
  Arms: Education by unpersonalised DVD
Behavioral: Standard care — standard care
  Arms: Standard Care
Behavioral: Education by DVD and dietician — Information on detrimental conseqences of hyperphosphatemia is presented on DVD and individual dietary counseling is given by dieticican
  Arms: Education by DVD and dietician

SUMMARY:
Hyperphosphatemia is a common and severe complication in chronic kidney disease patients treated with hemodialysis. A phosphate restricted diet and oral phosphate binders are the cornerstones in the prevention and treatment of this complication. However, noncompliance is an prevalent problem resulting in poorly controled hyperphosphatemia in a substantial proportion of hemodialysis patients. The present study aims at identifying risk factors for non compliance and also test the hypothesis that compliance can be improved by education patients on the consequences of hyperphosphatemia and the importance of diet and phosphate binder therapy.

ELIGIBILITY:
Inclusion Criteria:

* prevalent (>3months) hemodialysis patients
* aged > 18 years
* informed consent

Exclusion Criteria:

* decreased consciousness
* unstable
* medical contraindication for phosphorus restricted diet or phsophate binder therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
compliance | baseline and after intervention
  impact of education (by DVD and interview with dietician)on compliance with phosphorus restricted diet and phosphate binder therapy
serum phosphate levels | baseline and after intervention
  impact of education (by DVD and interview with dietician) on serum phosphate levels

SECONDARY OUTCOMES:
risk factors of noncompliance | baseline
  identification of risk factors for non compliance with emphasis on cognitive function and depression

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium